CLINICAL TRIAL: NCT00098397
Title: A Phase II Study Of Single Agent Depsipeptide (FK228) In Breast Cancer
Brief Title: FR901228 in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02641; MDA-2003-0895; N01CM17003 (NIH); CDR0000404163 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — romidepsin

ARMS (1):
- Treatment (romidepsin) (Experimental): Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: romidepsin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase II trial is studying how well FR901228 works in treating patients with metastatic breast cancer. Drugs used in chemotherapy, such as FR901228, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. FR901228 may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy and safety of FR901228 (depsipeptide) in patients with metastatic breast cancer.

SECONDARY OBJECTIVES:

I. Determine the clinical activity of this drug, in terms of progression-free survival, in these patients.

OUTLINE: This is a multicenter study.

Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 2.4-12.3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer

  * Metastatic disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
  * The following are not considered measurable disease:

    * Bone disease only
    * Pleural effusion
    * Peritoneal effusion
* Must have received prior anthracycline (doxorubicin or epirubicin) and/or taxane (paclitaxel or docetaxel) as adjuvant therapy or for advanced disease

  * Therapy with high-dose regimens or bone marrow transplantation is considered 1 prior regimen
* No known brain metastases
* Hormone receptor status:

  * Not specified
* Male or female
* Performance status - ECOG 0-1
* Performance status - Karnofsky 70-100%
* More than 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* AST or ALT ≤ 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance ≥ 60 mL/min
* QTc < 500 msec
* No New York Heart Association class III or IV congestive heart failure
* No myocardial infarction within the past year
* No uncontrolled dysrhythmia
* No poorly controlled angina
* No other significant cardiac disease
* No history of serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to FR901228
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No concurrent biologic agents
* No more than 1 prior chemotherapy regimen for metastatic disease
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior FR901228 (depsipeptide)
* No other concurrent chemotherapy
* Prior hormonal therapy for metastatic disease or as adjuvant therapy allowed
* More than 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy
* More than 2 weeks since prior minor surgery and recovered
* More than 4 weeks since prior major surgery and recovered
* Concurrent bisphosphonates allowed provided therapy was initiated ≥ 3 months ago
* No concurrent agents that cause QTc prolongation
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent drugs known to have histone deacetylase activity (e.g., valproic acid)
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-02; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Efficacy (complete and partial response) according to RECIST | Up to 14 months
Progression-free survival | From the first day of treatment to the first observation of disease progression or death due to any cause, assessed up to 14 months

SECONDARY OUTCOMES:
Toxicity as measured by the standard WHO grading system | Up to 14 months after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Cristofanilli, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States